SHEET OF INFORMATION FOR PARTICIPANTS IN

**RESEARCH STUDIES WITH SAMPLES** 

Study Title: EFFECT OF REGULAR CONSUMPTION OF HYDROXYTYROSOL

ON GLYCEMIC AND CHOLESTEROLEMIC METABOLISM IN HUMANS

Principal Investigator, Service/Unit, and Center: Dr. Ángeles Velasco Soria,

Family and Community Medicine, Mu-San Andrés Health Center

Promoter/Financier: Catholic University of San Antonio of Murcia/Fundación

Séneca

Version Number and Date: 01/03/2022, version 1.

INTRODUCTION

Considering the cardiovascular pathology risk you present, we are contacting you

to inform you about a study in which you are invited to participate. Our intention

is to provide you with correct and sufficient information so that you can evaluate

and decide whether or not to participate in this study. Before deciding whether to

participate or not, we kindly ask you to carefully read this document, which

includes information about this project. You can ask any questions that arise and

request clarification on any aspect of it. We will clarify any doubts that may arise

at any time. Additionally, you may consult with whomever you deem appropriate.

The project has the favorable report of an accredited Research Ethics Committee

in Spain.

**VOLUNTARY PARTICIPATION** 

You should know that your participation is voluntary, and you can decide not to

participate or change your decision and withdraw your consent at any time,

without altering your relationship with your doctor or causing any harm to your

treatment.

PURPOSE AND PROCEDURES OF THE STUDY:

1. What it consists of and its purpose: We aim to analyze the effect of

regular consumption of hydroxytyrosol on your cardiovascular system.

You will benefit from intensive monitoring over the next 2 and a half

months.

2. How it is carried out: If you consent to participate in the study, you will

be asked to consume 4 xylitol candies/day enriched with hydroxytyrosol

(60 mg/day) for 28 days, then rest for two weeks, and after that, you will

be asked to resume consuming 4 xylitol candies/day for another 28 days.

You will be scheduled a total of four times throughout the study for

peripheral blood extractions and to respond to dietary surveys. The

extractions pose no risk to the individual.

3. **Effects it will produce:** Hydroxytyrosol has been widely marketed as an

active compound for its potent antioxidant and anti-inflammatory effects,

so it can only provide beneficial effects for your health.

PROCEDURES FOR OBTAINING SAMPLES, DISCOMFORT, AND POSSIBLE

RISKS:

Some of the samples are obtained during the usual monitoring of your disease or

condition; others are requested because they are necessary to fulfill the

objectives of this study. Below, we explain what they are and the risks associated

with the procedures used to obtain them:

Blood samples: 4 blood samples will be obtained, and the amount extracted in

each analysis will be 10 mL of blood (2 EDTA vacutainers and 1 serum

vacutainer). For most people, needle punctures for blood extraction pose no

problem. However, occasionally, they can cause bleeding, bruising, discomfort,

infections, and/or pain at the blood extraction site. You may also feel dizzy. The

samples and associated data will be kept under appropriate security conditions,

and it is guaranteed that subjects cannot be identified through means considered

reasonable by individuals other than those authorized.

Additional data or samples may be necessary. In that case, your doctor will

contact you again to request your collaboration. You will be informed of the

reasons, and your consent will be requested again (see yes/no option at the end

of the sheet).

**EXPECTED BENEFITS:** 

No direct benefit from participating in the study is expected. However, the

knowledge gained from studies conducted using your samples and many others

can contribute to medical advancement and, therefore, to other people. You will

not receive any financial benefit from donating the samples and providing the

data, nor will you have rights over any commercial benefits from the discoveries

that may result from the research conducted.

**ANALYSIS SITE AND STORAGE OF SAMPLES:** 

During the study's development, your samples may be analyzed in various

laboratories and will be stored for 6 months, in anticipation of the need to repeat

any additional analysis related to the study's objectives. During this process, the

project's investigator/promoter will be responsible for the samples. They will be

used for measuring plasma markers of cardiovascular status, after which they will

be destroyed.

INFORMATION ON THE DESTINATION OF SAMPLES AND FUTURE USE

The extracted blood will be used for the measurement of biochemical parameters

(lipid profile, renal profile, hepatic profile, and basal glycemia) and a complete

blood count. The third vacutainer (EDTA) will be centrifuged at 3500 rpm, 15 mins,

at room temperature for plasma extraction. This plasma will be used for the

analysis of plasma markers using ELISA techniques (adiponectin, leptin, LDL-ox,

ghrelin, IL-6, PCR, and insulin). This plasma will be stored at UCAM at -80° for a

maximum period of 6 months. After the ELISAs are completed, the excess plasma

will be destroyed.

RIGHT TO WITHDRAW CONSENT

If you change your mind regarding the donation of biological samples and the

provision of the provided data, you have the right to request their destruction or

anonymization, through your doctor/investigator/principal investigator of the

collection/biobank. However, you should know that the data obtained in the

analyses conducted up to that point may be used for the requested purposes and

may be retained in compliance with the corresponding legal obligations.

CONFIDENTIALITY/PROTECTION OF PERSONAL DATA

Your samples will be coded, associating them with a code that cannot be related

to you. Only authorized personnel defined as researchers of this project will be

able to relate the information derived from the analyses carried out to information

about your identity.

This study is fully subject to Organic Law 3/2018 of December 5, on the Protection

of Personal Data and guarantee of digital rights, and Regulation (EU) 2016/679

of the European Parliament and of the Council of April 27, 2016, on Data

Protection (GDPR). Therefore, it is important that you know the following

information:

• Your personal data will be processed for the purpose indicated in the

signing document and will be kept for the necessary years to comply with

applicable current regulations.

• The Data Controller is the University Clinical Hospital "Virgen de la

Arrixaca" (Health Area I of Murcia/West), whose **Data Protection** 

Delegate (DPD) is Ms. Elena García Quiñones with address at Servicio

Murciano de Salud, C./ Central nº 7, Edificio Habitamia I, 30100,

Espinardo-Murcia (email: <a href="mailto:dpd-sms@carm.es">dpd-sms@carm.es</a>).

• The legal basis legitimizing the processing is your consent.

• Applicable regulations: Regulation (EU) No 536/2014 of the European

Parliament and of the Council of 16 April 2014 on clinical trials on medicinal

products for human use, and repealing Directive 2001/20/EC; Organic Law

3/2018, of December 5, on the Protection of Personal Data and guarantee

of digital rights, Law 14/2007, of July 3, on Biomedical Research; Royal

Legislative Decree 1/2015, of July 24, approving the consolidated text of

the Law on Guarantees and Rational Use of Medicines and Medical

Devices; Law 44/2003, of November 21, on the regulation of health

professions, as well as Law 14/1986, of April 25, on General Health, Law

41/2002, of November 14, on patient autonomy, and other current

legislation on health matters.

Your data will not be transferred, except in cases required by law or in

cases of medical emergency. However, you may revoke the consent given

at any time and exercise your rights of access, rectification, erasure,

objection, restriction of processing, and portability, to the extent

applicable, through written communication to the Data Controller as

follows, specifying your request, along with your ID card or equivalent

document:

- Principal Investigator of the study: Ángeles Velasco Soria

- Address: Family and Community Medicine Service of Mu-San Andrés

Health Center

Likewise, we inform you of the possibility of filing a complaint with the

Spanish Data Protection Agency (C/Jorge Juan, 6 Madrid 28001)

www.agpd.es

Access to your personal information will be restricted to the study

physician/collaborators, Health Authorities for inspection purposes, the Clinical

Research Ethics Committee, when necessary to verify the study's data and

procedures, but always maintaining their confidentiality.

The data collected for the study will be identified by a code, so that no information

that could identify you is included, and only your study physician/collaborators will

be able to relate this data to you and your medical history.

Based on this data, scientific communications may be prepared to be presented

at congresses or scientific journals, always maintaining the confidentiality of your

personal data.

You are informed that, in accordance with the provisions of the seventeenth

additional provision of Organic Law 3/2018, of December 5, on the Protection of

Personal Data and guarantee of digital rights, as well as Article 89 of Regulation

(EU) 2016/679, if your data are processed for research purposes in public health

and, in particular, biomedical research, the following will be carried out:

An impact assessment will be carried out to determine the risks arising

from the processing in the cases provided for in Article 35 of Regulation

(EU) 2016/679 or those established by the supervisory authority. This

assessment will specifically include the risks of re-identification linked to

anonymization or pseudonymization of data.

Scientific research will be subject to quality standards and, where

appropriate, international guidelines on good clinical practice.

Measures will be adopted, where appropriate, aimed at ensuring that

researchers do not have access to data identifying the data subjects. In

the event that this separation between data and the researcher cannot be

guaranteed, an express commitment to confidentiality by the researcher

will be guaranteed, as well as not to carry out any re-identification activity.

Specific security measures will be adopted to prevent re-identification and

unauthorized access by third parties.

IMPLICATIONS OF THE INFORMATION OBTAINED BY ANALYZING THE

SAMPLES

If you request it, you may be provided with information about the research studies

in which your samples have been used, as well as the general results of this

study.

If this study obtains data that may be clinically or genetically relevant to you, and

of interest to your health or that of your family, you may request that it be

communicated to you by your trial doctor if indicated in the box at the end of this

document. However, if the patient has indicated their refusal and when this

information, according to the responsible physician's criteria, is necessary to

prevent serious harm to their health or that of their biological relatives, a close

family member or representative will be informed, following consultation with the

center's Ethical Assistance Committee. The communication of this information will

be carried out by professionals who can adequately explain its relevance and the

options that may arise. In the case of clinically relevant genetic information, you

may receive the required genetic counseling.

In the case of a minor donor, upon reaching the age of majority, they will have the

right to receive this information and to revoke consent. If they do not exercise it,

it will be considered that the current document remains valid.

| biological sample is not used in certain research. | | | | | |
|---|---|---|---|---|---|
| If you wish t | to establish any re<br><b>indicate</b> | estrictions rega | arding the fu | uture use of t | he samples, |
| FUTURE R | ESEADOU | | | | |
| FUTURE RI | ESEARCH | | | | |
| | the possible reuse<br>ical areas related | • | data for res | earch purpos | es in health |

Discuss with your doctor the possibility of establishing restrictions so that your

## **INFORMED CONSENT FORM**

| | et Title:<br>OXYTYROS<br>BOLISM IN | | | REGUI<br>EMIC | | CONSUMPTI<br>CHOLESTE | |
|---|---|---|---|---|---|---|---|
| | | gator, Servio | | | | Ángeles Vela<br>h Center | asco Soria |
| | <b>oter/Financ</b><br>/Fundación | ` | icable):( | Catholic | Univer | sity of San | Antonio o |
| Partici | pant/Patient | t Information | | | | | |
| Name | | | | | | | |
| Investi | gator or Pe | rson Providir | ng Informa | tion | | | |
| Name | | | | | | | |
| | Sheet, whice | ch I attest w | vith my sig<br>erein. | gnature | as evid | ontent of this I | consent to |
| | that I can re | equest the revexplanations, | vocation o | f this co | nsent at | d free, and I used any time, with my present ar | nout having |
| | | • | | | | information de<br>e to my healtl | |
| □Y | ES | □NO | Phone | | or | email | contact |
| | | · · | | • | | ples and asso | |

Area I Murcia Oeste Madrid-Cartagena Road, s/n. El Palmar. 30120-Murcia T: 968 369 500

sheet:

| □YES □NO | O | | | | |
|---|---|---|---|---|---|
| | ent to be cor<br>al samples ar | ntacted in case<br>re needed: | additional i | nformation o | or additiona |
| □YES | □NO | Phone | or | email | contact |
| | | · | | | |
| Date: | | Pa | rticipant's/Pa | tient's Signa | ture |
| Date: | Invest | igator's or Pers | on Providing | Information' | s Signature |
| REVOCATION | OF CONSE | NT | | | |
| I, Mr./Ms | | | _, revoke the | e consent giv | ven on date |
| and I do not wi | sh to continu | e participating | in the study " | EFFECT OF | REGULAR |
| CONSUMPTIC | N OF | HYDROXYTYF | ROSOL ON | N GLYCE | MIC AND |
| CHOLESTERO | DLEMIC MET | ABOLISM IN H | UMANS." | | |
| Patient's Signa | ture: | | | | |
| Investigator's S | Signature: Da | te: | | | |

HOJA DE INFORMACIÓN PARA PARTICIPANTES EN ESTUDIOS DE INVESTIGACIÓN CON

**MUESTRAS** 

Titulo del estudio: EFECTO DEL CONSUMO REGULAR DE HIDROXITIROSOL

SOBRE EL METABOLISMO

GLUCÍDICO Y COLESTEROLEMICO EN HUMANOS

Investigador Principal, servicio/unidad y centro: Dra. Ángeles Velasco Soria,

Medicina Familiar y Comunitaria, Centro de Salud Mu-San Andrés

Promotor/financiador: Universidad Católica San Antonio de

Murcia/Fundación Séneca. № de versión y fecha: 01/03/2022,

versión 1.

INTRODUCCIÓN

Considerando el riesgo de patología cardiovascular que usted presenta, nos

dirigimos a usted para informarle sobre un estudio en el que se le invita a

participar. Nuestra intención es que reciba la información correcta y suficiente

para que pueda evaluar y juzgar si quiere o no participar en este estudio. Antes

de decidir si quiere participar o no, le rogamos lea detenidamente este

documento que incluye la información sobre este proyecto. Puede formular todas

las preguntas que le surjan y solicitar cualquier aclaración sobre cualquier

aspecto del mismo. Nosotros le aclararemos las dudas que puedan surgir en

cualquier momento. Además, puede consultar con las personas que considere

oportuno.

El proyecto cuenta con el informe favorable de un Comité de Ética de la

Investigación acreditado en España.

PARTICIPACIÓN VOLUNTARIA

Debe saber que su participación es voluntaria y que puede decidir no participar

o cambiar su decisión y retirar el consentimiento en cualquier momento, sin que

por ello se altere la relación con su médico ni se produzca perjuicio alguno en su

tratamiento.

PROPÓSITO Y PROCEDIMIENTOS DEL ESTUDIO:

<u>1-</u> <u>En qué consiste y para qué sirve:</u> nos proponemos analizar el efecto del consumo regular del hidroxitirosol sobre su sistema cardiovascular. **Usted se** 

beneficiará de un seguimiento intensivo durante los próximos 2 meses y medio.

<u>2-</u> <u>Cómo se realiza:</u> si usted consiente su participación en el estudio se le pedirá consumir 4 caramelos/día enriquecidos en hidroxitirosol (60 mg/día)

durante 28 días, descansará dos semanas y tras ello, se le pedirá volver a consumir 4 caramelos/día durante otros 28 días. Se le citará un total de cuatro

veces a lo largo del estudio para las extracciones de sangre periférica y responder a

**encuestas alimentarias.** Las extracciones no suponen ningún riesgo para el individuo.

<u>Qué efectos le producirá:</u> el hidroxitirosol se ha comercializado ampliamente

como compuesto activo por sus potentes efectos antioxidantes y antiinflamatorios, por lo que sólo puede aportar efectos beneficiosos para su

salud.

PROCEDIMIENTOS DE OBTENCIÓN DE MUESTRAS, MOLESTIAS Y

**POSIBLES RIESGOS:** 

Algunas de las muestras se obtienen durante el seguimiento habitual de su

enfermedad o proceso; otras son solicitadas porque son necesarias para cumplir

con los objetivos de este estudio. A continuación le explicamos cuáles son y los

riesgos asociados a los procedimientos utilizados para su obtención:

Muestras de sangre: se obtendrán 4 muestras de sangre y la cantidad extraída en

cada análisis será de 7 ml (1 vacutainer de EDTA y 1 vacutainer de suero) de

sangre. Para la mayoría de las personas, las punciones con agujas para la

extracción de sangre no suponen ningún problema. Sin embargo, en ocasiones,

pueden provocar hemorragias, hematomas, molestias, infecciones y/o dolor en

el punto de extracción de sangre. También puede sentirse mareado.

Las muestras y los datos asociados se mantendrán bajo las condiciones de

seguridad adecuadas y se garantiza que los sujetos no podrán ser identificados

a través de medios considerados razonables por personas distintas a las

autorizadas.

Es posible que sea necesario algún dato o muestras adicionales. En ese caso,

su médico se pondrá en contacto con usted para solicitarle de nuevo su

colaboración. Se le informará de los motivos y se le solicitará de nuevo su

consentimiento (ver opción sí/no al final de la hoja).

**BENEFICIOS ESPERADOS:** 

No se espera un beneficio directo por su participación en el estudio. No obstante,

los conocimientos obtenidos gracias a los estudios llevados a cabo a partir de

sus muestras y de muchas otras pueden ayudar al avance médico y, por ello, a

otras personas. No percibirá ningún beneficio económico por la donación de las

muestras y la cesión de los datos proporcionados, ni tendrá derechos sobre

posibles beneficios comerciales de los descubrimientos que puedan conseguirse

como resultado de la investigación efectuada.

LUGAR DE ANÁLISIS Y ALMACENAMIENTO DE LAS MUESTRAS:

Durante el desarrollo del estudio sus muestras pueden ser analizadas en

diversos laboratorios y se mantendrán almacenadas durante 6 meses, en

previsión de que fuera necesario repetir algún análisis adicional relacionado con

los objetivos del estudio. Durante este proceso el responsable de las muestras

será el investigador/promotor del proyecto. Serán utilizadas para la medida de

marcadores plasmáticos del estado cardiovascular tras lo cual serán destruidas.

INFORMACIÓN SOBRE EL DESTINO DE LAS MUESTRAS Y USO

**FUTURO** 

La sangre extraída será utilizada para la medida de parámetros bioquímicos

(perfil lipídico, perfil renal y hepático, glucemia basal, HOMA e insulina). El

vacutainer de EDTA se centrifugará a 3500 rpm, 15 mins, a temperatura ambiente

para la extracción de plasma. Ese plasma será utilizado para la medida de

marcadores plasmáticos mediante técnicas de ELISA (adiponectina, leptina,

LDL-ox, grelina). Ese plasma será centrifugado y almacenado en la UCAM a -

80º durante un plazo máximo de 6 meses. Al finalizar los ELISAs, el excedente

de plasma será destruído.

DERECHO DE REVOCACIÓN DEL CONSENTIMIENTO

Si cambiara de opinión en relación con la donación de las muestras biológicas y

la cesión de los datos proporcionados, tiene derecho a solicitar su destrucción o

anonimización, a través de su médico/investigador/investigador principal de la

colección/ biobanco. No obstante, debe saber que los datos que se hayan

obtenido en los análisis realizados hasta ese momento podrán ser utilizados para

los fines solicitados y podrán conservarse en cumplimiento de las obligaciones

legales correspondientes.

CONFIDENCIALIDAD/PROTECCIÓN DE DATOS PERSONALES:

Sus muestras estarán codificadas, asociándolas a un código con el que no será

posible relacionarle a usted con ellas. Sólo personal autorizado definido como

investigadores de este proyecto podrá relacionar la información derivada de los

análisis realizados con información sobre su identidad.

A este estudio les son plenamente de aplicación la Ley Orgánica 3/2018 de 5 de

diciembre, de Protección de datos de carácter Personal y garantía de los

derechos digitales y el Reglamento (UE) 2016/679 del Parlamento europeo y del

Consejo de 27 de abril de 2016 de Protección de Datos (RGPD). Por ello, es

importante que conozca la siguiente información:

Sus datos personales serán tratados con la finalidad indicada en el

documento objeto de firma y serán conservados durante los años

necesarios para cumplir con la normativa vigente aplicable.

• El Responsable del Tratamiento es el Hospital Clínico Universitario

"Virgen de la Arrixaca" (Área I de Salud-Murcia/Oeste), cuyo **Delegada de Protección de Datos** (DPD) es Doña **Elena García Quiñones** con dirección en Servicio Murciano de Salud, C./ Central nº 7, Edificio Habitamia I, 30100.

Espinardo-Murcia (correo electrónico: dpd-sms@carm.es).

La base jurídica que legitima el tratamiento es su consentimiento

, , ,

 Normativa aplicable: Reglamento (UE) n 536/2014 del Parlamento Europeo y del Consejo, de 16 de abril de 2014, sobre los ensayos clínicos de medicamentos

de uso humano, y por el que se deroga la Directiva 2001/20/CE; Ley Orgánica 3/2018, de 5 de diciembre, de Protección de Datos de Carácter Personal y

Garantía de los Derechos Digitales, Ley 14/2007, de 3 de julio, de Investigación biomédica; Real Decreto Legislativo 1/2015, de 24 de julio, por el que se aprueba el texto refundido de la Ley de garantías y uso racional de los medicamentos y

productos sanitarios; Ley 44/Ley 44/2003, de 21 de noviembre, de ordenación de las profesiones sanitarias, así como la Ley 14/1986, de 25 de abril, General de

Sanidad, la Ley 41/2002, de 14 de noviembre, de autonomía del paciente, y demás legislación vigente en materia sanitaria.

Sus datos no serán cedidos, salvo en los casos obligados por Ley o en casos de urgencia médica. No obstante, en todo momento podrá revocar el consentimiento prestado, así como ejercer sus derechos de acceso, rectificación, supresión, oposición, limitación del tratamiento y portabilidad, en la medida que sean aplicables, a través de comunicación escrita al Responsable del Tratamiento de la siguiente manera concretando su solicitud, junto con su DNI o documento equivalente:

- Investigador Principal del estudio: Ángeles Velasco Soria

 Domicilio: Servicio de Medicina Familiar y Comunitaria del Centro de Salud Mu-San Andrés

 Asimismo, le informamos de la posibilidad de presentar una reclamación ante la Agencia Española de Protección de Datos (C/Jorge Juan, 6 Madrid 28001) <a href="https://www.agpd.es">www.agpd.es</a>

El acceso a su información personal quedará restringido al médico del estudio/colaboradores, Autoridades Sanitarias en materia de inspección, al Comité Ético de Investigación Clínica, cuando lo precisen para comprobar los datos y procedimientos del estudio, pero siempre manteniendo la confidencialidad de los mismos.

Los datos recogidos para el estudio estarán identificados mediante un código, de manera que no se incluya información que pueda identificarle, y sólo su médico del estudio/colaboradores podrá relacionar dichos datos con usted y con su historia clínica.

A partir de dichos datos se podrán elaborar comunicaciones científicas para ser presentadas a congresos o revistas científicas siempre manteniendo en todo momento la confidencialidad de sus datos de carácter personal.

Se le informa que de conformidad a lo previsto en la Disposición adicional decimoséptima de la Ley Orgánica 3/2018, de 5 de diciembre, de Protección de Datos de Carácter Personal y garantía de los derechos digitales, así como del artículo 89 del Reglamento (UE) 2016/679, en el caso que con sus datos se lleve a cabo un tratamiento con fines de investigación en salud pública y, en particular, biomédica se procederá a:

 Realizar una evaluación de impacto que determine los riesgos derivados del tratamiento en los supuestos previstos en el artículo 35 del Reglamento (UE) 2016/679 o en los establecidos por la autoridad de

control. Esta evaluación incluirá de modo específico los riesgos de reidentificación vinculados a la anonimización o seudonimización de los

datos.

• Someter la investigación científica a las normas de calidad y, en su caso,

a las directrices internacionales sobre buena práctica clínica.

 Adoptar, en su caso, medidas dirigidas a garantizar que los investigadores no acceden a datos de identificación de los interesados. En el supuesto

de que no pueda garantizarse esta separación entre los datos y el investigador, se le garantiza un compromiso expreso de confidencialidad

por parte del investigador así como de no realizar ninguna actividad de reidentificación. Se adoptarán medidas de seguridad específicas para

evitar la reidentificación y el acceso de terceros no autorizados.

IMPLICACIONES DE LA INFORMACIÓN OBTENIDA AL ANALIZAR LAS

**MUESTRAS** 

En el caso de que usted lo solicite, se le podrá facilitar información acerca de los

estudios de investigación en los que se hayan utilizado sus muestras, así como

de los resultados generales del presente estudio.

En el caso de que en este estudio se obtengan datos que pudieran ser clínica o

genéticamente relevantes para usted, e interesar a su salud o a la de su familia,

podrá solicitar que le sean comunicados por su médico del ensayo si así lo indica

en la casilla que aparece al final de este documento. No obstante, si el paciente

hubiera indicado su negativa y cuando esta información, según criterio del

médico responsable, sea necesaria para evitar un grave perjuicio para su salud

o la de sus familiares biológicos, se informará a un familiar próximo o a un

representante, previa consulta al Comité de Ética Asistencial del centro. La

comunicación de esta información se llevará a cabo por profesionales que le

podrán explicar adecuadamente su relevancia y las opciones que se pudieran

plantear. En caso de información genética clínicamente relevante podrá recibir el

preceptivo consejo genético.

En el caso de donante menor de edad, llegada la mayoría de edad tendrá derecho a recibir esta información y a la revocación del consentimiento. En caso de que no lo ejerza, se considerará que el actual documento sigue vigente.

Hable con su médico sobre la posibilidad de que pueda establecer restricciones para que su muestra biológica no sea utilizada en determinadas investigaciones.

Si desea establecer alguna restricción en relación al uso futuro de las muestras, indique por favor en este apartado

| cuales: | |
|---------|------|
| | <br> |

## **INVESTIGACIONES FUTURAS**

Autorizo la posible reutilización de datos personales con fines de investigación en materia de salud y biomédica para finalidades o áreas de investigación relacionadas con este estudio.

## HOJA DE CONSENTIMIENTO INFORMADO

Título del proyecto: EFECTO DEL CONSUMOREGULAR DE HIDROXITIROSO SOBRE EL METABOLISMO GLUCÍDICO Y COLESTEROLEMICO EN HUMANOS

Investigador Principal, servicio/unidad y centro: Dra. Ángeles Velasco Soria,

Medicina Familiar y Comunitaria,

Centro de Salud Mu-San Andrés

**Promotor/financiador (si aplica):** Universidad Católica San Antonio de Murcia/Fundación Séneca.

Datos del participante/paciente

\_\_\_\_\_

Investigador o persona que proporciona la información

## Nombre:

Nombre

- He leído, he sido informado y comprendo el contenido de la presente hoja de Información, lo que acredito con mi firma en prueba de mi consentimiento en todo lo que en ella se contiene.
- Entiendo que mi participación es voluntaria y gratuita y comprendo que puedo solicitar la revocación de este consentimiento en cualquier momento, sin tener que ofrecer explicaciones y sin que esto repercuta en mis cuidados médicos presentes y/o futuros.
- Deseo que el médico del estudio me comunique la información derivada de la investigación que pueda ser relevante y aplicable para mi salud o la de mis familiares:
  - SI NO Teléfono o e-mail de contacto.....
- Consiento al almacenamiento y uso de las muestras biológicas y de los datos asociados para futuras investigaciones en las condiciones explicadas en esta hoja de información.
  - SI NO
- Consiento a ser contactado en el caso de necesitar más información o muestras biológicas adicionales.
  - SI NO Teléfono o e-mail de contacto.....

Fecha: Firma del Participante/paciente

Fecha: Firma del Investigador o persona que proporciona la información

**REVOCACIÓN DEL CONSENTIMIENTO** 

Yo, D/Dña..... revoco el consentimiento prestado en fecha y no deseo continuar participando en el estudio "EFECTO DEL CONSUMO REGULAR DE HIDROXITIROSOL SOBRE EL METABOLISMO GLUCÍDICO Y COLESTEROLEMICO EN HUMANOS".

Firma del paciente:

Firma del investigador: Fecha: